

## STATISTICAL ANALYSIS PLAN

Safety, Tolerability and Acceptability of Long-Acting Cabotegravir (CAB LA) for the Prevention of HIV among Adolescent Males – A Sub-study of HPTN 083

**HPTN 083-01** 

**Effective Date:** [Date of latest signature]

**Version:** [2.0]

Confidential All proprietary rights reserved



## STATISTICAL ANALYSIS PLAN

| Protocol Name: | Safety, Tolerability and Acceptability of Long-Acting Cabotegravir (CAB LA) for the Prevention of HIV among Adolescent Males— A Sub-study of HPTN 083 |
|---|---|
| Protocol Number: HPTN 083-01 | |
| Author(s): | Brett Hanscom, Timothy Skalland, Xu (Amber) Guo, Yuqing Jiao |
| Version: | 2.0 |

| Author(s): | | |
|---|---|---|
| Brett Hanscom | See eTMF Signature<br>Manifest | See eTMF Signature<br>Manifest |
| Lead Statistician | Signature | Date: DD/MM/YYYY |
| | See eTMF Signature | See eTMF Signature |
| Xu (Amber) Guo | Manifest | Manifest |
| Statistical Research Associate | Signature | Date: DD/MM/YYYY |
| Approvals: | | |
| Zo | nghui Digitally signed Zonghui Hu -S | by |

Signature

Hu-S

Date: 2023.01.06

16:44:38 -05'00'

Confidential All proprietary rights reserved

NIAID Statistical Reviewer

Date: DD/MM/YYYY



## **TABLE OF CONTENTS**

| 1. | LIST OF ABBREVIATIONS AND ACRONYMS | 5 |
|---|---|---|
| 2. | INTRODUCTION | 7 |
| 2.1<br>2.2<br>2.3<br>2.4 | STUDY OBJECTIVES AND ENDPOINTS | 8<br>9 |
| 2.5 | | |
| 3. | GENERAL DATA ANALYSIS CONSIDERATIONS | |
| 3.1<br>3.2 | | 10<br>10 |
| 4. | INTERIM ANALYSIS AND DATA MONITORING COMMITTEE | |
| 5. | GENERAL ANALYSIS METHODS | |
| 6. | TRIAL PARTICIPANT DISPOSITION | |
| 6.1<br>6.2<br>6.3 | 2 TREATMENT EXPOSURE | 14 |
| 6.4 | | |
| 7. | PRIMARY ANALYSES | 15 |
| 8. | PRIMARY ANALYSES | 16 |
| 8 | TOLERABILITY ENDPOINT ANALYSIS ACCEPTABILITY ENDPOINT ANALYSIS 8.3.1 Completion of scheduled injections 8.3.2 Preferred method for HIV prevention | 17<br>17<br>17 |
| 9. | SAFETY ANALYSES | 18 |
| 9.1<br>9.2<br>9.3 | 2 LABORATORY EVALUATIONS | 18 |
| 10. | IMMUNOGENICITY ANALYSES | 18 |
| 11. | PHARMACOKINETIC ANALYSES | 18 |
| 12. | SECONDARY ANALYSES | 19 |
| 13 | CHANGE HISTORY | 21 |



| 14. APPENDIX A – ADVERSE EVENTS OF SPECIAL INTEREST | 22 |
|-----------------------------------------------------|----|
| 15. APPENDIX B – VARIABLE DEFINITIONS | 23 |
| 16. APPENDIX C – IMPUTATION OF MISSING DATES | 25 |





## 1. LIST OF ABBREVIATIONS AND ACRONYMS

| Term/Abbreviation | Definition Definition |
|---|---|
| ADaM | Analysis Dataset Model |
| AEs | Adverse Events |
| AESI | AEs of Special Interest |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| CAB LA | Long-Acting Cabotegravir |
| CABG | Coronary Artery Bypass Grafting |
| CASI | Computer Assisted Self Interview |
| CBC | Complete Blood Count |
| CMC | Clinical Management Committee |
| СРК | Creatine Phosphokinase |
| CRF | Case Report Forms |
| CV | Coefficient of Variation |
| DAIDS | Division of AIDS |
| EC | Ethics Committee |
| FDA | (US) Food and Drug Administration |
| GEE | Generalized Estimating Equations |
| HBsAg | Hepatitis B Virus Surface Antigen |
| HBV | Hepatitis B Virus |
| HDL | High Density Lipoprotein |
| IM | Intramuscular |
| loR | Investigator of Record |
| IRB | Institutional Review Board |
| ISR | Injection Site Reaction |
| IUS | Intrauterine System |
| LDL | Low Density Lipoprotein |
| МО | Medical Officer |
| NIAID | National Institute of Allergy and Infectious Diseases |
| NICHD | National Institute of Child Health and Human Development |
| OHRP | Office for Human Research Protections |
| PTCA | Percutaneous Transluminal Coronary Angioplasty |

Confidential All proprietary rights reserved




| SD | Standard Deviation |
|--------|------------------------------------------------|
| SMC | Safety Monitoring Committee |
| SPDSMP | Study Progress and Data Safety Monitoring Plan |
| STI | Sexually Transmitted Infection |
| Tbili | Total Bilirubin |
| ULN | Upper Limit of Normal |
| US | United States |
| WBC | White Blood Cell |
| WHO | World Health Organization |





#### 2. INTRODUCTION

This SAP is intended to describe the final primary and secondary analyses upon completion of HPTN083-01. Sections of the SCHARP SAP template had to be adapted here to reflect the distinct single-arm outcomes, as opposed to the more common multi-arm studies that the template was designed for. Key variable definitions are included in Appendix B.

### 2.1 General Design Considerations

HPTN083-01 is a phase IIB single arm trial designed to establish the minimum safety, tolerability and acceptability data needed to support the use of cabotegravir long-acting injection (CAB LA) in an adolescent population, potentially transforming the field of HIV prevention for young people. The study target population is sexually active, healthy male adolescents aged below 18 years. The study target is to enroll more than 50 participants with at least 50 participants receiving at least one injection. Participant recruitment will take approximately 12 months.

Study participation includes Step 1: a 5-week oral CAB 30mg QD safety lead-in followed by Step 2: a series of 5 intramuscular (IM) injections of 3 mL (600 mg) cabotegravir administered at 8-week intervals after a 4-week loading dose (injections at weeks 5, 9, 17, 25 & 33). Adherence support strategies (e.g., counseling, reminders, pill cases) will be included to support pill-taking during the first five weeks and to support retention during the injectable phase. A safety visit will follow each injection to ascertain pharmacokinetic-peak safety data, including injection site reactions. Step 3: A blood draw visit, the +8 Week Visit, will follow the week 33 injection to monitor CAB drug levels. All participants who have received at least one injection will be followed for 48 weeks after their last injection. Waning levels of cabotegravir (the PK tail) will be covered with locally sourced oral TENOFOVIR/EMTRICITABINE (TRADE NAME: TDF/FTC, TRUVADA®) for daily use for 48 weeks. In Step 3 participants may also chose to continue with 8-week dosing of injectable of CAB-LA for 48 weeks (5 additional injections beyond the initial 5 injections, administered at weeks +8. +16, 24, +32, +40, and +48.) Behavioral and acceptability data will be collected via computer-assisted self-interview (CASI). Total participant commitment for the entire study is up to 87 weeks, or approximately 1.5 years. We anticipate recruitment for the study will take approximately 12 months.

Participants who discontinue study product during Step 2 for any reason other than HIV infection or AE occurrence will be transitioned to open label TDF-FTC for 48 weeks.

There are in total three study sites:

- Adolescent and Young Adult Research at the Core Center (AYAR at CORE), Chicago, IL;
- St. Jude Children's Research Hospital CRS, Memphis, TN;
- Fenway Health CRS, Boston, MA.

Study is sponsored by Division of AIDS (DAIDS), United States (US) National Institute of Allergy and Infectious Diseases (NIAID), Eunice Kennedy Shriver National Institute of Child Health and Human

All proprietary rights reserved




Development (NICHD),US National Institutes of Health (NIH), IND number is 122,744. Protocol Chair is Sybil Hosek, PhD and Protocol Co-chair is Lynda Stranix-Chibanda, MBChB, MMED

### 2.2 Study Objectives and Endpoints

#### Primary objectives:

• To evaluate the safety, tolerability, and acceptability of CAB LA in healthy, HIV-uninfected male adolescents aged below 18 years.

#### Secondary objectives:

- To examine adherence to and timeliness of injections over time among adolescent participants provided CAB LA and information regarding its safety and efficacy.
- To examine patterns of sexual risk behavior over time among adolescent participants provided CAB LA and information regarding its safety and efficacy.
- To evaluate the safety of oral CAB during step 1 (oral phase) as well as all study products during the aggregate oral+injectable period for all enrolled participants. Additionally, we will include an intention to treat analysis for the primary safety endpoint.
- To characterize the pharmacokinetics of CAB LA
- Additional exploratory analyses will be done with the laboratory and clinical data, including resistance mutations

To achieve the primary and secondary objective, the planned primary and secondary endpoints are:

#### **Primary endpoints:**

Safety endpoint: Proportion of participants experiencing any Grade 2 or higher clinical adverse events (AEs) and laboratory abnormalities among participants who receive at least one injection of CAB LA. Laboratory abnormalities include grade 2 or above on tests include (CRF: Chemistry Panel, Fasting Lipid Test Results, Urinalysis, Hematology):

- Renal function: Creatinine, Creatinine clearance
- Hematology: Hemoglobin, Platelets, WBC, Neutrophils, Lymphocytes
- Liver function: Alkaline phosphatase, AST, ALT, Total bilirubin
- Electrolytes: Phosphorus, Calcium
- Other chemistries: CPK, Glucose, Amylase, Lipase,
- Urine test: Protein, Glucose
- Fasting Lipid Test Results: Total cholesterol, Triglycerides, LDL, HDL

Tolerability endpoint: Proportion of participants who receive at least 1 injection and who discontinue receiving injections prior to the full course of injections due to intolerability of injection, frequency of injections or burden of study procedures. Reasons for intolerability may include:

- Injection site reaction
- Participant refused further participation<sup>1</sup>
- Participant lost to follow-up
- Participant is unwilling or unable to comply with required study procedures
- Participant refused further study product use
- Participant unable to adhere to visit schedule



<sup>1</sup>Excluding cases in which reason for termination is unrelated to intolerability

Acceptability endpoints: Proportion of participants who complete all scheduled injections and proportion of participants who receive at least one injection who would consider using CAB LA for HIV prevention in the future. This endpoint will be evaluated using CASI questionnaires at the last injection visit (Step 2, week 33) for participants who do not have acceptability data at the Step 2, week 33 visit (either due to a change in when the questionnaire items were administered<sup>2</sup>, missed the final injection visit, or discontinue injections early) and continue to step 3, acceptability endpoints are evaluated during the follow up phase (step 3, week +12). The primary acceptability outcome is:

If you wanted to protect yourself from getting HIV, which of the following product(s) would you prefer to use?

- Prefer not using a product
- Condoms only
- Oral PrEP pills only
- Injectable PrEP only
- Condoms and oral PrEP pills together
- Condoms and injectable PrEP together
- Prefer not to answer

#### **Secondary endpoints:**

- Proportion of injection visits that occurred "on-time"
  - O The target visit window for the week 5 injection is 0-3 days after the Week 5 visit date (allowing for the injection occurring on a different day from the W5 visit) and is +/-3 days from the target injection date for all other injection visits. Visits happening within the target window are considered "on-time"
- Change from enrollment of self-reported sexual behavior (number of sexual partners, increased episodes of anal sex without a condom) during the study period
- Proportion of participants experiencing Grade 2 or higher clinical AEs and laboratory abnormalities in the oral phase and the aggregate over the entire study period
- Plasma CAB pharmacokinetics

#### 2.3 Randomization

There is no treatment randomization as this study is a single arm, open label trial.

#### 2.4 Blinding

Participants and site staff will be unblinded throughout the trial.

#### 2.5 Sample Size and Power

The sample size for this protocol (n=50) is the number of participants agreed upon by the industry sponsor and regulators in order to provide supplementary safety and behavioral data on adolescents in collaboration with the HPTN 083 and HPTN 084 adult trials. The goal of the safety evaluation for this study is to identify safety concerns associated with CAB LA.

All proprietary rights reserved



| Table 2. Width of 95% confidence interval | |
|---|---|
| for estimated proportion as a function of | |
| the true proportion, | the true proportion, assuming a sample size |
| of 50. | |
| True proportion Width of 95% CI | |
| 0.1 | $\pm 0.083$ |
| 0.2 | $\pm 0.11$ |
| 0.3 | $\pm 0.13$ |
| 0.4 | $\pm 0.14$ |
| 0.5 | $\pm 0.14$ |

Since each of the primary endpoints is a proportion, Table 2 shows the precision (confidence interval width) that will be obtained for each endpoint with a sample size of 50.

Recognizing that some participants will not reach the first injection visit and/or may not receive any study injections due to personal or clinical concerns, the study will continue to recruit participants until it is clear that at least 50 participants will progress to the injection phase. Experience in the parent study HPTN 083 suggests that only a small proportion of participants will fail to reach the injection stage, and it is expected that approximately 5-7 additional enrollees may be needed in order to reach 50 participants in the injection phase.

#### 3. GENERAL DATA ANALYSIS CONSIDERATIONS

#### 3.1 Analysis Set(s)

Primary and secondary analyses will be carried out among the following populations:

Screened Population: Includes all participants who were screened for potential enrollment.

Injection Population: Includes enrolled participants who receive at least one injection of CAB LA.

Safety Population: Includes enrolled participants who began step 1 (oral phase).

Enrolled Population: Includes all enrolled participants.

Seroconverter Population: Includes all enrolled participants who seroconverted during the study.

TDF/FTC Population: All enrolled participants who were provided TDF/FTC during the study.

#### 3.2 Statistical Analysis Issues

AEs will be tabulated using MedDRA preferred terms. The number and percentage of participants experiencing each specific AE (All AEs, Grade 2 or higher, and SAEs) will be tabulated by severity and by relationship to study product. For the calculations in these tables, each participant's AEs will be counted once as the maximum severity and relationship to study product. AEs leading to temporarily or



permanently stopping drug will also be summarized. Methods for imputation of missing dates are described in Appendix C

#### 4. INTERIM ANALYSIS AND DATA MONITORING COMMITTEE

See: Study progress, data, and safety data monitoring plan (SPDSMP) for a detailed description of the safety monitoring committee (SMC) report and data and safety monitoring board (DSMB) report for this study.

#### 5. GENERAL ANALYSIS METHODS

Within the single arm, all primary and secondary outcome proportions with 95% CIs will be calculated.

#### 6. TRIAL PARTICIPANT DISPOSITION

#### 6.1 Disposition of Participants

The study will recruit participants to ensure that at least 50 participants progress to the injection phase, therefore more than 50 participants will be screened and enrolled.



## **Consort Diagram**





#### <sup>1</sup>Conditions in Step 1 that could disqualify a participant from transitioning to Step 2 are as follows:

- Pill count suggestive of less than 50% adherence at the Week 4 visit
- Missed or delayed Week 4 visit
- Grade 2 ALT at week 4, or grade 3 and above ALT anytime in step 1
- Grade 3 AE that is related to study product anytime in step 1, excluding ALT & CPK
- Grade 4 AE anytime in step 1, excluding ALT & CPK
- Grade 3 and above CPK and < Grade 3 ALT
- At substantial risk of HIV infection and/or qualifies for oral PrEP by local guidelines
- Any HIV reactive/positive test

#### Participant enrollment inclusion and exclusion criteria (see study protocol)

#### A. Inclusion Criteria

- 1) Assigned male at birth (including MSM, TGW, and gender non-conforming people)
- 2) At enrollment, below 18 years of age
- 3) At enrollment, body weight  $\geq$  35 kg (77 lbs.)
- 4) Willing to provide written informed assent/consent for the study and/or able to obtain written parental/guardian informed consent
- 5) Self-reported sexual activity with a male in the past 12 months
- 6) In general, good health, as evidenced by the following laboratory values:
  - a. Non-reactive / negative HIV test results
  - b. Absolute neutrophil count > 799 cells/mm3
  - c. Platelet count  $\geq 100,000/\text{mm}3$
  - d. Hemoglobin > 11g/dL
  - e. Calculated creatinine clearance ≥ 60 mL/minute using the modified Schwartz equation (≤ grade 2)
  - f. Alanine aminotransferase (ALT) < 2.0 times the upper limit of normal (ULN) and total bilirubin (Tbili)  $\le$  2.5 x ULN
  - g. Hepatitis B virus (HBV) surface antigen (HBsAg) negative and accepts vaccination
  - h. HCV Antibody negative
- 7) Willing to undergo all required study procedures
- 8) If currently on PrEP from a non-study source, willing to stop said PrEP prior to enrollment and agree to switch to oral CAB for the lead-in period and CAB LA injections.

#### **B.** Exclusion Criteria

- 1) Co-enrollment in any other HIV interventional research study or other concurrent studies which may interfere with this study (as provided by self-report or other available documentation);
- 2) Past or current participation in HIV vaccine trial with exception for participants who can provide documentation of receipt of placebo;
- 3) Exclusively had sex with biological females in lifetime;
- 4) In the last 6 months (at the time of screening):
- active or planned use of any substance use which would, in the opinion of the site investigator, would hinder study participation (including herbal remedies), as described in the IB or listed in the SSP, and/or Protocol Section 4.4
- 5) Known history of clinically significant cardiovascular disease, as defined by history/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or



percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease;

- 6) Inflammatory skin conditions that compromise the safety of intramuscular (IM) injections;
- 7) Tattoo or other dermatological condition overlying the buttock region that may interfere with interpretation of injection site reactions;
- 8) Current or chronic history of liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy);
- 9) Known history of clinically significant bleeding;
- 10) Surgically-placed or injected buttock implants or fillers, per self-report. Contact the CMC for guidance regarding questions about individual cases
- 11) A history of seizure disorder, per self-report;
- 12) Medical, social or other condition that, in the opinion of the site investigator, would interfere with the conduct of the study or safety of the participant (e.g., provided by self-report, or found upon medical history and examination or in available medical records);
- 13) Plans to move out of the geographic area within the next 18 months or otherwise unable to participate in study visits, according to the site investigator.

#### 6.2 Treatment Exposure

During step 1 (oral phase) staff are required to observe participants take one pill at enrollment, week 2 and week 4. Pill counts will occur at visits for week 2 and 4.

All injections during step 2 (injection phase) will be administered (and therefore directly observed) by study staff. Injections will be considered "on-time" if they occur in the visit window, described in the secondary analyses (section 12).

Blood samples will be collected throughout the study from all participants and assayed for plasma CAB concentrations. PK sample times include pre-dose trough samples at W5, W9, W17, W25, and W33 (final concentration in injection phase), 1-week post injection samples at W6, W10, W18, W26, W34, with a final sample at +8-weeks following the final injection. For participants advancing to Step 3 and do not elect to continue with CAB injections, additional follow-up samples will be collected at +24, +36 and +48-weeks following the final injection and at the HIV confirmatory visit.

#### 6.3 Protocol Deviations

Protocol deviations will be summarized in regular reports to the SMC, the details of which are available in the SPDSMP. Serious protocol deviations may result in participants being terminated from the trial and/or being excluded from analyses. The decision to exclude participant data from the analyses will be made based on independent review. Deviations resulting in failure to progress to the injection phase would exclude such participants from the pertinent analysis datasets (except for the secondary safety analyses, which are limited to the oral phase only).



#### 6.4 Unplanned enrollment discontinuation

In January 2022 the HPTN leadership determined that the study accrual rate was insufficient to meet the target enrollment in a reasonable amount of time, and study enrollments were stopped after a total accrual of nine participants.

#### 7. BASELINE DATA

The following data will be described overall, and by site:

Demographics (Table 1):

- Age (continuous mean, SD, median, min max; categorical (≤16, > 16): n (%))
- Gender identity
- Race
- BMI
  - o Age standardized BMI z-score (continuous mean, SD, median, min max)
  - o Classification as obese, overweight, normal, thinness, severe thinness based on z-score
    - *Note: The Clinical Study Report will report BMI without the use of z-scores*
- Housing security\*
  - O Do you have a regular place or home where you stay and store your things? (yes/no)
- Food security\*
  - O In the past 6 months, how frequently did you worry that your household would not have enough food?

Sexual behaviors / HIV Risk Perception (Table 2):

During the past month the participant had\*:

- o a primary partner
- o transactional sex with male sex partners
- o # male and/or transgender female sex partners
- o # male and/or transgender female sex partners who are reported to be HIV positive
- o # episodes of receptive anal sex
- # episodes of receptive anal sex without condom
- o # episodes of receptive anal sex without condom, with HIV+ or unknown partner
- # episodes of insertive anal sex
- # episodes of insertive anal sex without condom
- o # episodes of insertive anal sex without condom, with HIV+ or unknown partner
- STIs present at enrollment:
  - o Gonorrhea
  - Trachomatis
  - Syphilis
- Hepatitis testing at screening/enrollment
  - o HBV
  - o HCV


All proprietary rights reserved



- HIV risk perception\*:
  - o How much do you personally feel at risk of getting infected with HIV?

#### *Mental health* (Table 3):

- Depression indices<sup>1</sup>
  - CES-D-10\* (continuous mean, SD, median, min max; categorical (≤10: not depressed,
     >10: depressed): n (%))
  - PHQ9 (continuous mean, SD, median, min max; categorical (none-minimal, mild, moderate, moderately severe, severe): n (%))
- Intimate partner violence (IPV)\*
  - o In the past 6 months, have any of your partners punched, slapped, kicked, bit you, or caused you any type of physical harm?
  - o In the past 6 months, have any of your partners insulted, ignored or humiliated you, yelled at you, or made you feel ashamed or bad about yourself?
  - o In the past 6 months, have any of your partners forced you to have sex or perform any sexual act, or touched you sexually in any way that you did not want?
  - o In the past 6 months, have any of your partners made you feel afraid, unsafe or in danger?
- Primary care post-traumatic stress disorder screening questionnaire (PC-PTSD-4)\* (continuous mean, SD, median, min max; categorical (≤2: no PTSD, >2: potential PTSD): n (%))
  - o Note: The Clinical Study Report will not include this summary of PC-PTSD-4
- alcohol/substance use\*
  - o How often do you have a drink containing alcohol?
  - o How often do you have six or more drinks on one occasion?
  - o In the past month, did you have a drink containing alcohol just before or during sex?
  - o In the past month, how often have you used each of the following substances?
    - Cannabis (Also called marijuana, pot, grass, dakka, dagga or hash)
    - Amphetamine-type stimulants (For example Tik/Crystal Meth, ecstasy, speed, or diet pills)
    - Prescription drugs for non-prescription purposes (For example codeine (including cough syrup), efavirenz, valium)

<sup>1</sup>Internal consistency of Depression Index summaries (addendum to Table 3):

- 1. Tabular cross-frequency of the categories for CES-D-10/PHQ9
- 2. Scatterplot of the values of either index, with color-coding based on whether they agree on qualitative risk of depression
  - a. Note: The internal consistency evaluations will not be included in the Clinical Study Report

#### 8. PRIMARY ANALYSES

For each of the three primary endpoints the number and proportion of participants will be computed along with corresponding 95% confidence intervals. Each summary will be provided both overall and by site. Endpoint descriptions are available in section 2.2.

<sup>\*</sup>CASI questionnaire variables



#### 8.1 Safety endpoint analysis

*Cohort*: Injection population

Analysis description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities (reported as adverse events) from the first injection visit to 8 weeks after the last Step 2 injection visit, or Week 41, whichever comes first. See Section 3.2 for details regarding aggregation and tabulation of AEs.

#### 8.2 Tolerability endpoint analysis

*Cohort*: Injection population

Analysis description: Number and percent of participants who receive at least 1 injection and who discontinue receiving injections prior to the full course of injections due to intolerability of injection or burden of study procedures. Reasons for intolerability may include:

- a. Injection site reaction
- b. Burden of study procedure
  - i. Participant refused further participation
  - ii. Participant is unwilling or unable to comply with required study procedures
  - iii. Participant refused further study product use
  - iv. Participant unable to adhere to visit schedule

#### 8.3 Acceptability endpoint analysis

#### 8.3.1 Completion of scheduled injections

Population: Injection population and Enrolled population

Analysis description: Number and percent of participants who complete all scheduled injections<sup>1</sup>

<sup>1</sup>Definition of completing all scheduled injections for participants who are confirmed HIV positive or discontinue product due to the following reasons:

- Death
- Early study closure
- HBV infection

#### During Step 1:

Enrolled population: completed all 0 of 0 scheduled injections Injection population: not applicable, did not receive injection

#### During Step 2:

Both enrolled and injection populations: completed all injections whose target window closed prior to death/seroconversion/product discontinuation date

#### 8.3.2 Preferred method for HIV prevention

Population: Injection population



Analysis description: Number and percent of participants who choose 'injectable PrEP' or 'condoms and injectable PrEP' when asked the question "If you wanted to protect yourself from getting HIV, which of the following product(s) would you prefer to use?"

#### 9. SAFETY ANALYSES

See section 8.1 above. In addition to the primary safety outcomes (grade 2 or higher), AEs and laboratory data will be summarized in the closed DSMB report (described in the SPDSMP).

#### 9.1 Adverse Events and Deaths

Adverse events of special interest (AESI) will be summarized in the Clinical Study Report. Planned AESI summaries for the CSR are described in Appendix A.

#### 9.2 Laboratory Evaluations

Population: Safety population

Description: Laboratory findings for CBC (hemoglobin, platelets, WBC, neutrophils, lymphocytes), chemistries (urea, creatinine, CPK, glucose, calcium, phosphorous, amylase, lipase), liver function (AST, ALT, total bilirubin, alkaline phosphatase) and fasting lipid profile (total cholesterol, triglycerides, HDL, LDL) will be reported by grade, as defined in the "Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events". The proportion of laboratory findings qualifying as Grade 2 or above will be presented. Baseline laboratory values will be summarized by site using: median, 1st and 3rd quartiles, and min and max. Change from baseline in laboratory values will be summarized at follow up visits using: median, and 1st and 3rd quartile. Summaries involving values and changes from baseline at scheduled visit time points will consider values from scheduled visits only, and in the case of missing values, results will not be carried forward from interim (unscheduled) visits. For summaries and analyses involving changes in laboratory values over time or maximum change from baseline (e.g. shift tables), values from interim (unscheduled) visits will also be considered.

#### 9.3 Other Safety Measures

#### 10. IMMUNOGENICITY ANALYSES

NA

#### 11. PHARMACOKINETIC ANALYSES

Plasma will be collected during Steps 1 and 2 for pharmacologic assessment of CAB concentrations. Plasma and DBS will also be collected in Step 3, and if a study participant seroconverts, for potential pharmacologic analysis of plasma TFV and DBS TFV-DP concentrations, respectively, to assess PrEP adherence, and for potential HIV genotyping. Analysis details are provided in the current version of the Pharmacokinetics Analysis Plan



#### 12. SECONDARY ANALYSES

For binary secondary endpoints, the number and proportion of endpoints will be computed along with corresponding 95% confidence intervals. Each summary will be provided both overall and by site. CSR analysis will be only summarized overall. Endpoint descriptions are available in section 2.2.

#### 12.1 Plasma CAB pharmacokinetics

Analysis details are provided in the current version of the Pharmacokinetics Analysis Plan

## 12.2 Proportion of participants experiencing Grade 2 or higher clinical AEs and laboratory abnormalities in the oral phase and over the entire study period

Cohort: Safety population

Analysis description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities from:

- 1. enrollment to week 5 (oral phase (step 1), including interim visits).
- 2. enrollment to 8 weeks following the last injection received (aggregate over oral+injection phases (step 1-step 2) including interim visits)

# 12.3 Proportion of participants receiving one or more injections who experience Grade 2 or higher clinical AEs and laboratory abnormalities from initial injection to 36 weeks later

Population: Injection population

Analysis description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities from the first injection visit to approximately 36 weeks later regardless of whether participants received all 5 injections. For participants receiving all 5 injections, the end date is 8 weeks following the week 33 injection visit. For participants discontinuing study product early and moving on to Step 3, the end date is 36 weeks after the initial injection. Participants who terminate early are included in the analysis and censored at the date of termination.

#### 12.4 Proportion of injection visits that occurred "on-time"

Population: Injection population

Analysis description: Number and percent of injection visits (up to 5 per participant) that occur "on-time", using the number of injections given as the denominator. This will be presented along with the total number and percent of injections given, among all intended injections (i.e. 5 injections per participant).

<sup>1</sup>The target injection date is defined by the W5 visit i.e. for the initial injection, the target injection date is 0 days (same day), and is +28, +84, +140, +196 days from the W5 visit for injections 2-5, respectively. The target visit window for injection visits for the week 5 injection is 0 to 3 days after the W5 visit (if the injection could not be done on the same day as the W5 visit), for all other injection visits (W9, W17, W25, W33) the target window is +/-3 days from the target injection date. Injection dates happening within the target window are considered "on-time".



# 12.5 Change from enrollment of self-reported sexual behavior (number of sexual partners, and number of episodes of anal intercourse without a condom) during the study period

Note: This secondary analysis will not be included in the Clinical Study Report.

Population: Enrolled population

*Analysis description*: Counts of sexual partners and episodes of anal intercourse without a condom will be summarized (mean and median) at enrollment and each regular Step 1 and Step 2 follow-up visit (W4, W5, W9, W17, W25, W33, +8).

## 12.6 Evaluate rates of HIV drug resistance among participants who acquire HIV infection during the study

Population: Seroconverter population

*Analysis description*: Data from steps 1, 2, and 3 will be included. The number of cases of drug resistance will be summarized. All cases of drug resistance among incident HIV infections will be described.



### 13 CHANGE HISTORY

| Ve | rsion | Affected | Activity Description |
|---|---|---|---|
| Number | Effective<br>Date | Section(s) | |
| 1.0 | 02/20/2021 | All sections | First version of SAP was developed. |
| 2.0 | Date of<br>last<br>signature | 2, 3, 6, 7-9,<br>11, 12, 13,<br>16, 17 | Revisions based on new option to continue CAB injections during Step 3. Added study populations and definitions. Updated consort diagram, primary and secondary outcomes/analyses, including addition of secondary outcome 12.6. Updated acceptability endpoint definition, and reference to PK analysis plan. Additional details to account for changes to schedule of visits and data collection, due to new CAB option in Step 3. Added sections: 13 (ad hoc analysis), appendices A, B and C (AEs of special interest, variable definitions and imputation of missing data). Most revisions are designed to harmonize with HPTN 084-01 SAP 3.0. |



### 14. APPENDIX A - Adverse Events of Special Interest

Adverse events of special interest (AESI) have been determined for CAB based on pre-clinical and clinical experience, along with information for the integrase inhibitor class of HIV medications safety profile. These are adverse events for which more detailed summaries of event characteristics are of interest.

The identification and classification of AESI will be based on MedDRA preferred terms as specified in the ADRG (Analysis Data Reviewers Guide). The current MedDRA version used for the preferred terms in the ADRG is v25.1. Preferred terms will be updated in the ADRG if a new version becomes available before the database lock.

Table 1 below shows the adverse events of special interest identified and reasons for including.

Table 1 Adverse Events of Special Interest (Clinical Study Report only)

| AESI | Product Implicated | Reason for Including as AESI |
|---|---|---|
| Hepatic Safety Profile: Assessment of risk of hepatoxicity | CAB | Clinical, Class, Regulatory<br>Interest, |
| Hypersensitivity Reactions (HSR) | CAB | Class, Regulatory Interest, |
| Rash | CAB | Class, Regulatory Interest |
| Neuropsychiatric Events | CAB | Clinical, Class, Regulatory<br>Interest, |
| Injection Site Reactions (ISR) | CAB | Clinical, Regulatory Interest |
| Seizures and Seizure-like events | CAB | Clinical, Regulatory Interest |
| Weight Gain | CAB | Clinical, Class, Regulatory<br>Interest |
| Rhabdomyolysis | CAB | Clinical, Class, Regulatory<br>Interest |
| Pancreatitis | CAB | Clinical, Therapeutic Area,<br>Regulatory Interest |
| Impact on Creatinine | CAB | Regulatory Interest,<br>Therapeutic Area |


All proprietary rights reserved

#### HPTN083-01 Statistical Analysis Plan 17 Jan 2023 | SCHARP-TMF-32741 | 2.0



| Hyperglycemia/new onset diabetes mellitus CAB Observation from 083, Class | Hyperglycemia/new onset diabetes mellitus | CAB | Observation from 083, Class |
|---|---|---|---|
|---|---|---|---|

Common ISR adverse events are defined by MedDRA preferred terms including injection site pain, injection site induration, injection site nodules and preferred terms of any other ISR exceeding the threshold as specified in the ADRG. ISRs will be explored regardless of IP relationship.

Each one of the AESIs described in Table 3 will be explored via the data listings in more detail. Listings will summarize Adverse events that occurred during Step 1 and/or Step 2 of the study and will contain information to assess the following.

**Event Characteristics:** The characteristics of all event occurrences during the post-baseline period will look at event characteristics (serious, drug-related, leading to withdrawal, or Grade 3/4, fatal), number of events per participant, outcome, maximum grade or intensity and action taken.

**Time to First Event (TTFE) and Duration of Events:** Time of onset and duration of event will be provided.

In addition, Pyrexia Plus includes PT: (Chills – 10008531, Feeling of Body Temperature Change - 10061458, Feeling Hot - 10016334, Body Temperature Increased - 10005911, Pyrexia - 10037660, Influenza Like Illness - 10022004, Fever – 10016558) events will be looked at in relation to timing of previous injection.

No formal summaries or statistical comparisons are planned for AESI.

#### 15. APPENDIX B - Variable Definitions

#### 1. CES-D-10 (score/categories)

Create a score based on 10 items below (in CASI questionnaire):

In the list below, please indicate how often you have felt this way during the past week by ticking the appropriate box for each question:

- 1. I was bothered by things that usually don't bother me.
- 2. I had trouble keeping my mind on what I was doing.
- 3. I felt depressed.
- 4. I felt that everything I did was an effort.
- 5. I felt hopeful about the future.
- 6. I felt fearful or afraid.
- 7. My sleep was restless.
- 8. I was happy.
- 9. I felt lonely.
- 10. I could not "get going", I did not feel motivated.

#### **Scoring:**

| - 2 | | | | |
|---|---|---|---|---|
| | Rarely or none of the | Some or a little of the | Occasionally or a moderate | All of the time |
| | time (less than 1 day) | time (1-2 days) | amount of time (3-4 days) | (5-7 days) |


All proprietary rights reserved




| Questions 5 & 8 | 3 | 2 | 1 | 0 |
|---------------------|---|---|---|---|
| All other questions | 0 | 1 | 2 | 3 |

The total score is calculated by finding the sum of 10 items. Score as 'missing' if 1 or more items are missing/prefer not to answer. Any score  $\geq$ 10 is considered depressed.

#### 2. PHQ-9 (score/categories)

Create a score based on values from 9 questions (Not at all = 0, Several days = 1, More than half the days = 2, Nearly every day = 3):

Over the last 2 weeks, how often have you been bothered by the following problems?

- 1. Little interest or pleasure in doing things
- 2. Feeling down, depressed, or hopeless
- 3. Trouble falling or staying asleep, or sleeping too much
- 4. Feeling tired or having little energy
- 5. Poor appetite or overeating
- 6. Feeling bad about yourself or that you are a failure or have let yourself or your family down",
- 7. Trouble concentrating on things, such as reading the newspaper or watching television",
- 8. Moving or speaking so slowly that other people could have noticed. Or the opposite being so fidgety or restless that you have been moving around a lot more than usual
- 9. Thoughts that you would be better off dead, or of hurting yourself

PHQ-9 score obtained by adding score for each question (total points). Score as 'missing' if 1 or more items are missing. Then categories of depression severity are created from the total score according to: 0-4: None-minimal, 5-9: Mild, 10-14: Moderate, 15-19: Moderately Severe 20 - 27: Severe.

#### 3. PC-PTSD-4 (score/categories)

Create a score based on values from 4 questions (yes = 1, no = 0):

In your life, have you ever had any experience that was so frightening, horrible, or upsetting that, in the past month, you:

- 1. Have had nightmares about it or thought about it when you did not want to?
- 2. Tried hard not to think about it or went out of your way to avoid situations that reminded you of it?
- 3. Were constantly on guard, watchful, or easily frightened?
- 4. Felt empty, numb or detached from others, activities, or your surroundings?

If missing or prefer not to answer any questions, then code score as missing. For non-missing scores, a score of 0-2 fails to indicate PTSD, and  $\geq$  3 indicates the potential for PTSD, which can be determined by a clinical interview.


All proprietary rights reserved 



#### 4. Age-standardized BMI z-score

Based on World Health Organization (WHO) tool:

(1) <a href="https://www.who.int/tools/growth-reference-data-for-5to19-years/indicators/bmi-for-age">https://www.who.int/tools/growth-reference-data-for-5to19-years/indicators/bmi-for-age</a>.

With instructions for calculations (see section "Computation of centiles and z-scores", link to pdf: "instructions in English"):

(2) <u>https://cdn.who.int/media/docs/default-source/child-growth/growth-reference-5-19-years/computation.pdf?sfvrsn=c2ff6a95\_4</u>

Age-specific values of necessary parameters L(t), M(t), and S(t) can be downloaded from the website (1) (see section: "Expanded tables for constructing national health cards" link to dataset "z-scores: girls")

Categorical BMI classification based on age-standardized BMI z-score as follows:

- Obesity: >+2
- Overweight: >+1 and <+2
- Normal: >-2 and  $\leq$ +1
- Thinness: >-3 and  $\leq$ -2
- Severe thinness: ≤-3

#### 16. APPENDIX C – Imputation of missing dates

#### Missing Start and Stop Dates for Prior and Concomitant Medication, and Medical History

The Assumption is to consider the most conservative judgment when imputing.

#### Start date:

When imputing a start date ensure that the new imputed date is sensible i.e. is prior to the end date and the general rules are:

- 1. If start date is completely missing, start date will not be imputed
- 2. If year and month are present and day is missing, set day to the 1st day of month.
- 3. If year and day are present and month is missing, then set month to January.
- 4. If year is present and month and day are missing, set month and day to January 1st.

#### Stop date:

- 1. If end date is completely missing, end date will not be imputed
- 2. If year and month are present and day is missing, set day to the last day of month.
- 3. If year and day are present and month is missing, set month to December
- 4. If year is present and month and day are missing, set month and day to December 31st.

#### Missing Start and Stop Dates for Adverse Events (including ISRs)



The Assumption is to consider the most conservative judgment when imputing.

#### Start date:

- 1. If start date is completely missing, start date is set to date of first dose.
- 2. If (year is present, and month and day are missing) or (year and day are present, and month is missing):
  - a. If year = year of first dose, then set month and day to month and day of first dose.
  - b. If year < year of first dose, then set month and day to December 31st.
  - c. If year > year of first dose, then set month and day to January 1st.
- 3. If month and year are present and day is missing:
  - a. If year = year of first dose and
    - i. If month = month of first dose, then set day to day of first dose date.
    - ii. If month < month of first dose, then set day to last day of month.
    - iii. If month > month of first dose, then set day to 1st day of month.
  - b. If year < year of first dose, then set day to last day of month.
  - c. If year > year of first dose, then set day to 1st day of month.

#### Stop date:

If the outcome of the AE was ongoing or unknown, then the rules outlined below will not be applied.

- 1. If stop date is completely missing, stop date is set to date of study discontinuation.
- 2. If (year is present, and month and day are missing) or (year and day are present, and month is missing):
  - a. If year = year of study discontinuation, then set month and day to month and day of study discontinuation.
  - b. If year < year of study discontinuation, then set month and day to December 31st.
  - c. If year > year of study discontinuation, then set month and day to December 31st.
- 3. If month and year are present and day is missing:
  - a. If year = year of study discontinuation and
    - i. If month = month of study discontinuation, then set day to day of study discontinuation date
    - ii. If month < month of study discontinuation, then set day to last day of month.
    - iii. If month > month of study discontinuation, then set day to last day of month.
  - b. If year < year of study discontinuation, then set day to last day of month.
  - c. If year > year of study discontinuation, then set day to last day of month.

#### Missing Start and Stop Dates for Protocol Deviations

The Assumption is to consider the most conservative judgment when imputing.

#### Start date:

When imputing a start date ensure that the new imputed date is sensible i.e. is prior to the end date and the general rules are:

- 1. If start date is completely missing, start date will not be imputed
- 2. If (year is present, and month and day are missing) or (year and day are present, and month is missing), set month and day to January 1st.
- 3. If year and month are present and day is missing, set day to the 1st day of month.



#### Stop date:

- 1. If end date is completely missing, end date will not be imputed
- 2. If (year is present, and month and day are missing) or (year and day are present, and month is missing), set month and day to December 31st.
- 3. If year and month are present and day is missing, set day to the last day of month.



## Signature Page for SCHARP-TMF-32741 v2.0

| Reason for signing: Approved | Name: Xu Guo<br>Role: Data Analytics<br>Date of signature: 17-Jan-2023 19:54:18 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: Brett Hanscom<br>Role: Hutch SDMC<br>Date of signature: 17-Jan-2023 23:02:14 GMT+0000 |

Signature Page for SCHARP-TMF-32741 v2.0